CLINICAL TRIAL: NCT03295422
Title: Investigator Initiated Randomized Controlled Trial Comparing Two Radiofrequency Ablation Strategies in Patients With Persistent Atrial Fibrillation
Brief Title: Comparison of Two Pulmonary Vein Ablation Techniques for Persistent AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sequoia Hospital (Other)
Responsible Party: Principal Investigator, Christopher E. Woods, MD, PhD, Study Principal Investigator, Sequoia Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Persistent AF Study 01
Record Dates: First submitted 2017-09-24; First posted 2017-09-27 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Chronic Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Radiofrequency ablation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RF ablation PVI alone (Active Comparator): RF catheter ablation of pulmonary veins alone
  Interventions: Procedure: RF ablation PVI alone
- RF ablation PVI plus LPAW (Experimental): RF catheter ablation PVI plus left atrial posterior wall
  Interventions: Procedure: RF ablation PVI plus LPAW

INTERVENTIONS:
Procedure: RF ablation PVI alone — A series of RF applications will be delivered around both sets of pulmonary veins with complete entry and exit block obtained around the antrums of all 4 pulmonary veins.
  Other Names: Catheter ablation of the pulmonary veins
  Arms: RF ablation PVI alone
Procedure: RF ablation PVI plus LPAW — A series of RF applications will be delivered around both sets of pulmonary veins with complete entry and exit block obtained around the antrums of all 4 pulmonary veins. In addition, a roof and posterior line will be placed in the left atrium to achieve entrance and exit block on the posterior wall. Entry block will be confirmed by placing a circular mapping catheter in multiple locations along the posterior wall and confirming lack of presence of any local potentials. Exit block will be confirmed on the posterior wall with pacing at 10 amps from the ablation catheter at multiple locations within the box as well as all lines.
  Other Names: Catheter ablation of the pulmonary veins plus posterior wall
  Arms: RF ablation PVI plus LPAW

SUMMARY:
Investigator initiated, randomized controlled trial of two radiofrequency (RF)ablation protocols currently performed in the electrophysiology lab, but have not been studied prospectively to identify which, if either technique, is superior for individuals with persistent atrial fibrillation (AF). Two-hundred subjects will be consecutively enrolled and randomized to either pulmonary vein isolation only or pulmonary vein isolation plus posterior left atrial wall isolation

DETAILED DESCRIPTION:
Atrial fibrillation, the most common type of cardiac arrhythmia in clinical practice, affects approximately 2.7 million U.S. adults. Percutaneous catheter ablation is an effective treatment option for individuals with persistent AF. Pulmonary vein isolation (PVI) has emerged as the gold standard for paroxysmal AF with excellent success rates, however, individuals with persistent AF procedural efficacy from pulmonary vein isolation is not optimal. Therefore, improved ablation strategies for these individuals are needed.

This randomized controlled trial will compare two radiofrequency ablation strategies, PVI alone and pulmonary vein isolation plus left posterior atrial wall (LPAW) isolation in individuals with persistent AF. Both strategies are currently used to treat persistent AF, but no randomized controlled trial ahs been conducted to investigate which strategy is more efficacious.

Two-hundred subjects will be randomized into groups of 50 to undergo a radiofrequency ablation procedure for AF. For group 1, a series of radiofrequency applications will be delivered around both sets of pulmonary veins. For group 2, a series of radiofrequency applications will be delivered around both sets of pulmonary veins and along a roof and low posterior line of the left atrial wall.

All subjects will be followed at 1 month, 3 months, 6 months, and 1 year post ablation. If indicated, antiarrhythmic drugs will be discontinued. For the first month, subjects will receive a continuously recording electrocardiogram heart card to monitor for AF, and then two-week ambulatory monitors at 3 months and one year post ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Have symptomatic persistent AF (i.e., a sustained episode lasting more than 7 days).
2. Refractory to at least one antiarrhythmic agent.
3. Undergoing ablation for the first time.

Exclusion Criteria:

1. Paroxysmal AF
2. Sustained atrial fibrillation lasting more than 3 years
3. Left atrial diameter of 60 mm or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year freedom from recurrent atrial arrhythmias | 1 Year
  The primary hypotheses that PVI+PI will lead to a greater percentage of patients free from atrial arrhythmias after single ablation procedures than PVI alone.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Woods, MD, PhD, Principal Investigator — Dignity Health, Sequoia Hospital
Locations (1):
- Dignity Health, Sequoia Hospital, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT03295422/Prot_001.pdf